CLINICAL TRIAL: NCT03315000
Title: The Effect of Vilanterol Against Methacholine-induced Bronchoconstriction in Mild Asthmatics
Brief Title: Effect of Vilanterol on Methacholine Challenge Results
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, Department of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VIL-2017
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: methacholine; airway hyperresponsiveness
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — vilanterol; fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vilanterol (Experimental): Vilanterol (25mcg)+ fluticasone (100mcg) inhaled through Ellipta® inhaler
  Interventions: Drug: Vilanterol and Fluticasone Furoate
- Fluticasone (Experimental): Fluticasone (100mcg) monotherapy inhaled through Ellipta® inhaler
  Interventions: Drug: Fluticasone Furoate
- Placebo (Placebo Comparator): Lactose powder inhaled through Ellipta® inhaler
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Vilanterol and Fluticasone Furoate — Same as vilanterol arm description
  Other Names: Breo
  Arms: Vilanterol
Drug: Fluticasone Furoate — Same as fluticasone arm description
  Other Names: Arnuity
  Arms: Fluticasone
Drug: Placebos — Same as placebo arm description
  Other Names: lactose powder
  Arms: Placebo

SUMMARY:
The study will assess the degree of bronchoprotection provided by the ultra long-acting beta2 agonist vilanterol against methacholine-induced bronchoconstriction.

DETAILED DESCRIPTION:
This will be a double-blind, three-way crossover study comparing combination vilanterol+fluticasone with fluticasone monotherapy and a placebo (vilanterol is not available as a monotherapy). The order in which the treatments are given will be randomized and each treatment will be separated by a minimum one-week washout. Fifteen asthmatic participants will be recruited from the local community. Methacholine challenge testing (MCT) with the two-minute tidal breathing protocol will be used to quantify the bronchoprotective effects (if any) of each treatment against methacholine-induced bronchoconstriction.

Each participant will undergo a total of nine methacholine challenges. After a baseline methacholine challenge, the randomized treatment (identity unknown to investigator or participant) will be administered through an Ellipta® (multi-dose dry powder inhaler). Thirty minutes following treatment administration, a second methacholine challenge will be performed. At 24 hours post-treatment, each participant must re-visit the lab for one methacholine challenge. The same process will be followed for each treatment.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 or older
* stable mild-to-moderate asthma
* baseline methacholine PC20 less than or equal to 8mg/mL
* FEV1 greater than or equal to 65% of predicted

Exclusion Criteria:

* Use of long-acting anticholinergic or long-acting beta2 agonist within 30 days of study
* pregnant or nursing
* diabetes
* hypokalemia
* cardiovascular, prostate, kidney, or urinary retention problems
* lactose-intolerant
* allergy-induced asthma symptoms or upper respiratory tract infection within four weeks of study
* current smokers
* past smokers with smoking history >10 pack years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline methacholine PC20 (bronchoprotection) at 30 min post-treatment | baseline versus 30 min post-treatment
  assessed by dose shift of geometric mean methacholine PC20 data

SECONDARY OUTCOMES:
Change from baseline methacholine PC20 (bronchoprotection) at 24 hours post-treatment | baseline versus 24 hours post-treatment
  assessed by dose shift of geometric mean methacholine PC20 data

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Journal Publication

REFERENCES:
- [Derived] Westbury GLM, Blais CM, Davis BE, Cockcroft DW. Bronchoprotective effect of vilanterol against methacholine-induced bronchoconstriction in mild asthmatics: A randomized three-way crossover study. Ann Allergy Asthma Immunol. 2018 Sep;121(3):328-332. doi: 10.1016/j.anai.2018.07.005. Epub 2018 Jul 12. PMID 30017826